CLINICAL TRIAL: NCT04090294
Title: Assessment of Early Outcomes of Roflumilast in Patients With Non Cystic Fibrosis Bronchiectasis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Ahmed Abd El-Gawad Mohamed Okash, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Roflumilast in bronchiectasis
Record Dates: First submitted 2019-08-21; First posted 2019-09-16 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Roflumilast

STUDY DESIGN:
Intervention Model Description: 35 patients will receive roflumilast for three months and improvement regarding performance , frequency of exacerbation and pulmonary function test will be assessed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Roflumilast -non roflumilast (Experimental): 35 patients will receive Roflumilast for three months and improvement regarding dyspnea scales , Pulmonary function Test , Six minutes walking test and bronchectasis severity index (FACED) score pre and post therapy will be assessed.
  patients will receive Roflumilast 500 Mcg. Tablet Once daily for Three months and then base line assessment will be repeated to evaluate improvement.
  Interventions: Drug: Roflumilast

INTERVENTIONS:
Drug: Roflumilast — Roflumilast is a phosphodiesterase (PDE) type 4 inhibitor will be prescribed for three month for the study group. the patients will then be assessed for improvement regarding exacerbation frequency , performance and pulmonary function test.
  patients will receive Roflumilast 500 Mcg. Tablet once daily for three months
  Other Names: phosphodiestrase 4 inhibitor (PDE4)

SUMMARY:
Aim of the work

Assessment of early outcome of using Roflumilast in patients with bronchiectasis regarding:

* Severity of symptoms
* Frequency of exacerbations
* Change in pulmonary function
* Systemic inflammation

DETAILED DESCRIPTION:
Bronchiectasis is defined by the presence of permanent and abnormal dilation of the bronchi. This usually occurs in the context of chronic airway infection causing inflammation. The main clinical manifestation is a productive cough. Bronchiectasis is currently nearly always diagnosed using high-resolution computed tomography (HRCT) scanning. The main diagnostic features are: 1) internal diameter of a bronchus is wider than its adjacent pulmonary artery; 2) failure of the bronchi to taper; and 3) visualization of bronchi in the outer 1-2 cm of the lung fields.

* From a series of benzamide derivatives, roflumilast (3-cyclo-propylmethoxy-4-difluoromethoxy-N-[3,5-di-chloropyrid-4-yl]-benzamide) was identified as a potent and selective PDE4 inhibitor. It inhibits PDE4 activity from human neutrophils. PDE4 inhibitors were demonstrated to inhibit inflammatory cytokine and mediator release from inflammatory cells. In addition, it inhibits neutrophil chemotaxis or migratory activity. Lastly, PDE4 inhibitor promotes apoptosis of these cells .
* Studies have demonstrated the efficacy of roflumilast in patients with both asthma and COPD, where roflumilast improved lung function and reduced exacerbation rates.
* Bronchiectasis is a chronic destructive lung disease, which is characterised by persistent bacterial colonization, bronchial inflammation, reduced mucociliaryclearance, and in some patients progressive tissue damage. There is evidence of an associated influx of neutrophils into the lungs of these patients , resulting in the expectoration of large volumes of purulent sputum containing neutrophils and their products, so In patients with bronchiectasis, there is also neutrophilic inflammation as in COPD.

  * The PDE4 inhibitor, roflumilast, was evaluated in short term clinical trial of non-cystic fibrosis bronchiectasis. It has been shown symptomatic improvement from baseline Park J. found that 16 weeks Roflumilast treatment in patients with non cystic fibrosis bronchiectasis significantly reduce CAT score and improve the symptoms of non-CF bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above, male or female.
* Non / Ex-smokers.
* Confirmed diagnosis of bronchiectasis based on high-resolution computed tomography scan.
* Significant sputum production (≥ 10 ml per day).

Exclusion Criteria:

* Non-stable patients who need ICU admission /mechanical ventilation.
* Active smokers.
* Moderate to severe liver impairment (Child-Pugh B or C) and/or sever renal impairment (c. clearance less than 30ml/min).
* Known psychiatric illness
* Concomitant use of strong cytochrome P450 inducers (e.g. rifampicin)
* Patients who are hypersensitive to roflumilast.
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of efficacy of Roflumlilast regarding control of patients with non cystic fibrosis bronchiectasis | 3months . outcomes will be evaluated after 1month and at the end of the study (3months).
  Assessment of efficacy of Roflumilast on severity of symptoms in patients with bronchiectasis. Frequency of Exacerbation in the three months assessment and need of hospitalization will be the main parameter for efficacy of the new treatment described as number/ 3 months
Assessment of efficacy of roflumlilast in change of performance in patients with non cystic fibrosis bronchiectasis | 3months . outcomes will be evaluated after 1month and at the end of the study (3months).
  Assessment of efficacy of roflumilast on change dyspnea scale namely mMRCP evaluated at the start of the study and after 1 month and 3 months
Assessment of efficacy of roflumlilast on change in Pulmonary function in patients with non cystic fibrosis bronchiectasis | 3months . outcomes will be evaluated after 1month and at the end of the study (3months).
  Assessment of efficacy of roflumilast on change in pulmonary function test in patients with bronchiectasis regarding : change in FEV1 by liter per second
Assessment of efficacy of roflumlilast on change of symptoms in patients with non cystic fibrosis bronchiectasis | 3months . outcomes will be evaluated after 1month and at the end of the study (3months).
  Assessment of efficacy of roflumlilast on severity of symptoms in patients with bronchiactasis evaluated by bronchectasis severity index (FACED) score.
Assessment of efficancy of roflumlilast on change in systemic inflammation in patients with non cystic fibrosis bronchiectasis | 3months . outcomes will be evaluated after 1 month and at the end of the study (3 months).
  Assessment of efficacy of roflumlilast on systemic inflammation in patients with bronchiectasis regarding CRP by mg per L

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Shaddad, Lecturer, Principal Investigator — Assuit University - Assuit - Egypt

IPD SHARING:
Plan to Share IPD: Yes
the investigator group is welling to share all Data after finishing the study
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 24 Months
Access Criteria: open Access

REFERENCES:
- [Background] Sousa LP, Lopes F, Silva DM, Tavares LP, Vieira AT, Rezende BM, Carmo AF, Russo RC, Garcia CC, Bonjardim CA, Alessandri AL, Rossi AG, Pinho V, Teixeira MM. PDE4 inhibition drives resolution of neutrophilic inflammation by inducing apoptosis in a PKA-PI3K/Akt-dependent and NF-kappaB-independent manner. J Leukoc Biol. 2010 May;87(5):895-904. doi: 10.1189/jlb.0809540. Epub 2010 Jan 26. PMID 20103769
- [Background] Barker AF. Bronchiectasis. N Engl J Med. 2002 May 2;346(18):1383-93. doi: 10.1056/NEJMra012519. No abstract available. PMID 11986413
- [Background] Grootendorst DC, Gauw SA, Verhoosel RM, Sterk PJ, Hospers JJ, Bredenbroker D, Bethke TD, Hiemstra PS, Rabe KF. Reduction in sputum neutrophil and eosinophil numbers by the PDE4 inhibitor roflumilast in patients with COPD. Thorax. 2007 Dec;62(12):1081-7. doi: 10.1136/thx.2006.075937. Epub 2007 Jun 15. PMID 17573446
- [Background] van Schalkwyk E, Strydom K, Williams Z, Venter L, Leichtl S, Schmid-Wirlitsch C, Bredenbroker D, Bardin PG. Roflumilast, an oral, once-daily phosphodiesterase 4 inhibitor, attenuates allergen-induced asthmatic reactions. J Allergy Clin Immunol. 2005 Aug;116(2):292-8. doi: 10.1016/j.jaci.2005.04.023. PMID 16083782
- See also: 2. King PT, Holdsworth SR, Freezer NJ, Villanueva E, Holmes PW. Characterisation of the onset and presenting clinical features of adult bronchiectasis. Respir Med. 2006;100:2183-2189. [PubMed] [Google Scholar] — http://www.ncbi.nlm.nih.gov/pubmed/16650970
- See also: The preclinical pharmacology of roflumilast--a selective, oral phosphodiesterase 4 inhibitor in development for chronic obstructive pulmonary disease.Pulm Pharmacol Ther 2010;23:235-56. 10.1016/j.pupt.201 — https://doi.org/10.1016/j.pupt.2010.03.011